CLINICAL TRIAL: NCT05403606
Title: "Guarantee Assessment in Skin Prevention Adapted to Real Life With a Connected Device After a Spinal Cord Injury."
Acronym: GASPARD-SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC21_0044
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; pressure ulcer; prevention; medical advice; visual feedback
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (GASPARD®) (Experimental): Spinal cord injured patient with the connected electronic seat pressure measurement device (GASPARD®), a traditional follow-up and having received therapeutic education at the end of the treatment
  Interventions: Device: GASPARD®
- Control group: (No Intervention): Spinal cord injured patient with traditional follow-up with therapeutic education at discharge from initial care

INTERVENTIONS:
Device: GASPARD® — Spinal cord injured patient with the connected electronic seat pressure measurement device (GASPARD®), a traditional follow-up and having received therapeutic education at the end of the treatment
  Arms: Experimental Group (GASPARD®)

SUMMARY:
The investigators propose to test an embedded device on the seat of the wheelchair of paraplegic or tetraplegic patients (Gaspard), allowing on the one hand the continuous measurement of the pressures of seat, on the other hand a retro-control connected to the cell phone of the participants to inform them on these variables of seat (bad positioning, prolonged supports etc...) This study will be carried out over a long period of time (1 year), in an ergonomic situation of integration in the daily life of the participants. The main objective of this randomized controlled study is to study the difference in the incidence of pressure sores according to the use or not of this device. A qualitative study of the experience and perceived benefit of its use and a medico-economic study are associated to judge the expected interest in making this type of embedded device more systematically integrated into the classic movement equipment (wheelchair and seat cushion) of people with a spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with acquired spinal cord injury Traumatic or non-traumatic origin of the spinal cord injury

  * Motor level < C6
  * Complete or incomplete injury (AIS A, B and C impairment scale)
  * Primarily using a manual wheelchair (with or without electric propulsion assistance) as a means of mobility
  * At least 18 years of age
  * At any time after the occurrence of the spinal cord injury
  * Patients discharged from the center, with a first post-injury rehabilitation completed
  * Having participated in a specific therapeutic patient education on pressure ulcer prevention
  * No pelvic pressure sores under medical or surgical treatment at the time of inclusion
  * No aorto-iliac arterial disease that may promote pelvic ischemia (arterial Doppler <6 months)
  * Patient using a cushion approved by the HAS
  * Patients with a smartphone

Exclusion Criteria:

* Congenital spinal cord injury
* Motor level of the lesion > or = C6
* Incomplete motor lesion (AIS D and E)
* Patients who walk as their primary mode of ambulation
* Use of an electric wheelchair
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients per group for whom a pressure ulcer occurred. | 1 year

SECONDARY OUTCOMES:
Incremental cost-utility ratio of a connected electronic seat pressure measurement device (GASPARD®) compared to traditional management (= without device) | 1 year
Skin Risk Knowledge Questionnaire Revised-SMNAC (Skin Management Needs Assessment Checklist) | 1 year
Cross-analysis and thematic analysis of the comments made during the focus groups, particularly with regard to the perception of one's ability to take charge of one's health and the connected dimension of the device. | 1 year
Frequency of pelvic location of pressure ulcer (sacrum, ischium, trochanters). Frequency of pressure ulcer stages (1 to 4) | 1 year
Number of pressure sores per patient | 1 year
Analysis of Hospital Anxiety and Depression Scale (HADS) scores and International Pain Data Set variables. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MARC LE FORT, Principal Investigator — Nantes University Hospital; GAELLE AUDAT, Principal Investigator — CRRF l'Arche; RECH CELIA, Principal Investigator — Raymond Poincaré Hospital; KERDRAON Jacques, Principal Investigator — CRRF Kerpape; GELIS ANTHONY, Principal Investigator — Centre Mutualiste Neurologique Propora

IPD SHARING:
Plan to Share IPD: No